CLINICAL TRIAL: NCT04683419
Title: Modified Thoracoscopic Pleural Cryobiopsy in Diagnosis of Exudative Pleural Effusion of Undetermined Etiology
Brief Title: Modified Thoracoscopic Pleural Cryobiopsy in Diagnosis of Exudative Pleural Effusion
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Alexandria University (Other)
Responsible Party: Principal Investigator, Ayman Baess, Associate Professor, Alexandria University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 0105678
Record Dates: First submitted 2020-12-05; First posted 2020-12-24 (Actual); Last update posted 2020-12-24 (Actual); Status verified 2020-12

CONDITIONS: Pleural Effusion
Keywords: Thoracoscopy; Cryobiopsy
MeSH Terms: conditions — Pleural Effusion

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients with pleural effusion of Undetermined etiology (Experimental): Patients with undiagnosed exudative pleural effusion will undergo modified pleural cryobiopsies and conventional pleural forceps biopsies in the same settings
  Interventions: Device: Modified Thoracoscopic pleural Cryobiopsy

INTERVENTIONS:
Device: Modified Thoracoscopic pleural Cryobiopsy — Thoracoscopic pleural biopsy will be taken with a modified technique "raising of the parietal pleura by injection of saline, adrenaline and xylocaine, then taking the biopsy via a cryoprobe"

SUMMARY:
Background: Rigid thoracoscopy is the gold standard tool for diagnosing exudative pleural effusion but sometimes it is difficult to obtain sufficient biopsies using the conventional forceps.

Objectives: This study evaluated the efficacy, safety and diagnostic value of a modified technique using cryoprobe to obtain pleural biopsies during thoracoscopy.

Methods: This is a single center prospective study in patients who will undergo rigid thoracoscopy using conventional rigid forceps followed by a cryoprobe from the same site after injection of subpleural mixture of adrenaline and xylocaine. Biopsies will be reviewed by an independent pathologist; any complications will be recorded, and all patients will be followed up post procedure.

DETAILED DESCRIPTION:
Brief Summary: Background: Rigid thoracoscopy is the gold standard tool for diagnosing exudative pleural effusion but sometimes it is difficult to obtain sufficient biopsies using the conventional forceps..

Objectives: This study evaluated the efficacy, safety and diagnostic value of a modified technique using cryoprobe to obtain pleural biopsies during thoracoscopy.

Methods: This is a single center prospective study in patients who will undergo rigid thoracoscopy using conventional rigid forceps followed by a cryoprobe from the same site after injection of subpleural mixture of adrenaline and xylocaine. Biopsies will be reviewed by an independent pathologist and any complications will be recorded.

Detailed Description: The present study will prospectively enroll 24 patients with undiagnosed exudate pleural effusion who are admitted to Alexandria Main University Hospital , chest department .

All patients will undergo thoracoscopy whom biopsies will be taken using the modified cryo-biopsy technique and the conventional forceps biopsy technique.

All included patients will be subjected to :

* Full history .
* Clinical examination .
* Routine laboratory investigations including complete blood picture, prothrombin activity and international normalized ratio (INR).
* Radiological evaluation including:

  * Plain x-ray poster-anterior view,
  * Computed topography scan of the chest
  * Ultrasound examination of the pleural cavity.
* Thoracentesis and pleural fluid analysis will be done including:

  * Microbiological examination.
  * Biochemical examination (Protein-Glucose-LDH).
  * Cytopathological examination.
* Follow up chest x-ray will be done .

Thoracoscopy:

I. Endoscopy suite:

The endoscopy suite contains :

1. Thoracoscopy table: with a back that can be raised .
2. A separate sterile table for placing the thoracoscope, trocar, forceps and other accessories.
3. Adjustable aspiration equipment for the pleural fluid (BMI VAC60).
4. Simple anesthetic equipment with nasal prongs and central oxygen.
5. Mayo stand placed sideways across the thoracoscopy table to hold the instruments.
6. Electrocautery unit (ERBE ICC 200 EA, Germany).
7. Electrical systems which are attached to a voltage regulator and auxiliary electrical supply independent of the mains.
8. An included area for handwashing and area for sterilization of instruments.
9. Mobile carts for light sources and video camera.
10. Ultrasonography device (Philips ClearVue 350, Mexico)
11. Electronic medical records including Desktop computer, TV-Box (AV Grabber PRO WS-VR203P), and LCD screen (LG 32") .

II. Sterile conditions:

III. Patient monitoring during the procedure:

IV. Personnel:

The main personnel will be; a physician , an assistant operator , an assistant nurse, a circulating nurse outside the sterile field and a medical worker

V. Equipment:

A. Thoracoscope:

Rigid thoracoscope: (Karl Storz GmbH & Co., Germany) will be used .

Instruments for rigid thoracoscopy included:

* A metallic trocar with multifunctional valve with insufflation stopcock, 11mm in diameter and autoclavable.
* A 10 mm straight forward telescope 0º with angled eyepiece with a 6 mm working channel (26038AA, K. Storz-Endoskope, Tuttlingen, Germany)

B. Forceps:

Rotational biopsy forceps with connector pin for uni-polar coagulation will be used. They are 5 mm in diameter.

C. Cryo-Equipment:

The cryo-equipment consists of a cylinder containing cryogen stored under high pressure, a console (cryo-machine) that controls the flow of cryogen and a catheter with a cryoprobe at one end to freeze target tissue.The thoracoscopist will use a foot pedal to regulate the flow of the cryogen through the catheter from the cylinder to the cryoprobe. The cryo-machine available is ERBOCRYO CA, Tubingen, Germany.

D. Flexible Cryoprobe:

A flexible cryoprobe with a diameter of 2.4 mm was used to collect the pleura by firmly attaching it to the biopsy site for (10 - 30seconds) (ERBE, technikGmBH, Tubingen, Germany).

E. Rigid Cryoprobe:

A rigid cryoprobe will be used and the same steps were adopted as in case of using flexible Cryoprobe(ERBE, technikGmBH, Tubingen, Germany).

F. Transbronchial Needle:

A trans-bronchial needle with 1.8 mm diameter will be used to inject subpleural mixture of lidocaine 2%and epinephrine diluted by normal saline 9% to facilitate pleural biopsy using cryo technique (Aspiration needle ENDO-FLEX, Voerde, Germany).

VI. Phases of medical thoracoscopy :

A. Patient positioning:

The patient lay on the healthy side with the diseased side up , the arm will be raised over the head and a pillow will be placed on the table under the patient's flank to widen the targeted intercostal spaces.

B. Selecting the point of entry:

The point of entry will be determined near the mid-axillary line within the axillary triangle (bounded anteriorly by the inferior edge of pectoralis major muscle, posteriorly by the anterior edge of the latissimus dorsi muscle, cranially by the axillary apex and caudally down to the level of diaphragmatic insertion). The point of entry will be usually determined by ultrasonography and most commonly it is in the fifth, sixth or seventh intercostal spaces.

C. Anaesthesia:

Medical thoracoscopy in the current study will be done under local anaesthesia with moderate sedation . In some cases, general anesthesia will be applied if patients refuse local anesthesia and moderate sedation.

For local anaesthesia, the following steps will be done:

* The previously marked site of entry will be palpated with the index and middle fingers of one hand .
* Between the two fingers, a syringe (small bore, 27 gauge) will be filled with 1ml of 2% lidocaine (Debocaine®) will be used for intradermal injection to produce a small bleb.
* The local anaesthetic (10-15 ml of 2% lidocaine) in a larger bore syringe will infiltrate subcutaneously and in the intercostal muscles down to the parietal pleura.
* The path of the needle will be perpendicular to the chest wall ensuring that the needle has not penetrated a vascular structure.

At the location of the parietal pleural, about 8-10 ml of lidocaine will be infiltrated.The caudal rim of the upper rib will be infiltrated to anaesthetize the intercostal nerve as well as the periosteum of the rib itself then a further lidocaine depot of about 8-10 ml will be then injected around the cranial rim of the lower rib.

D. Performance of rigid thoracoscopy will be done using rigid scopes through single-port technique.

Steps performed:

* A 10-15 mm horizontal incision will be made at the pre-determined point of entry , parallel to and in the middle of the selected intercostal spaces
* Blunt dissection will be performed through the subcutaneous space, the intercostal muscles and the parietal pleura using a haemostat .
* Once the parietal pleura is opened, the index finger will be introduced through this opening to examine the pleura.
* The trocar is held with its head in the operator's palm and the extended index finger on its shaft in a position that limited the depth of insertion for safety's sake.
* The movement of air in and out of the pleural space should be heard during patient's respiration. Furthermore, pressure equilibrium with the atmosphere is established .
* The trocar will be removed, leaving the cannula in place then the pleural fluid will be aspirated by a suction catheter.
* The rigid scope will be then introduced through the cannula to gain access to the inside of the pleura.
* The pleural space will be visualized by the thoracoscope video-transmission.
* After removal of the pleural fluid, a systematic exploration of the chest cavity will be performed.
* In case of fine adhesions , mechanical separation will be possibly done using the forceps or the scope itself.
* In case of vascular adhesions or thick fibrous bands, electrocautery forceps will be used.

Biopsy techniques: thoracoscopic pleural biopsies are usually taken from the suspected parietal pleural lesions using the rigid forceps. They are taken against a rib to minimize the risk of vessel or nerve injury. Those biopsies will be taken using single-port single-instrument rigid technique .

Two techniques for the rigid forceps will be applied in the current study, first "punch biopsy" technique and second "strip biopsy" technique where the parietal pleura is grasped and gently pulled toward the operator then pulled sideways and in shearing motion, a "strip" of pleura could be isolated. In certain occasions, large "several centimeters long" specimens may be obtained .

Five to ten biopsies of suspicious pleural lesions will be taken. In cases of suspected malignancy , 10-12 parietal pleural biopsies from different locations will be taken.

Another biopsy technique will then be applied after subpleural injection of the diluted mixture of epinephrine and lidocaine 2% using transbronchial needle till subpleural raising and bleb is formed, then introduction of the cryoprobe (either the flexible or the rigid ) to be attached to the biopsy site then the operator uses the cryo-machine pedal for delivering the freezing effect through the cryoprobe for at least (10 - 30) seconds then grasping the cryoprobe with the attached pleural biopsy will be done, The tissue attached to the tip of the cryoprobe will be spontaneously thawed in normal saline at room temperature, three to five biopsies of suspicious pleural lesions were taken.

No biopsies will be taken from the anterior costoparietal pleura for fear of bleeding secondary to injury of the internal mammary artery .

Chest tube insertion:

The chest tube will be connected to a thoracic drainage device. chest x-ray will be then performed, and the patient will be discharged and scheduled for follow-up. Days till chest tube removal will be calculated and recorded.

VII. The follow-up of patients:

Follow up will be done following the procedure to detect any complications till discharge of the patient.

Follow-up will be carried out by chest x-ray.

VIII. Grading for Fat cells and crushed cells:

the measurement of the quantity of fat cells and crushed cells will be done as follows , if there will be no presence was marked as negative and if less than 5% of the biopsy will be marked as + and if 5-25% of the biopsy will be marked as ++ and if more than 25% it will take +++ in both limbs of the cryo and forceps techniques.

IX. Post-procedure complications Post-procedure complications will be recorded with the followings;

1. Local site ''wound'' infection.
2. Pneumothorax/ incomplete lung expansion.
3. Fever
4. Pain
5. Bleeding.

ELIGIBILITY:
Inclusion Criteria:

* Adult patient with undiagnosed exudative pleural effusion

Exclusion Criteria:

* Any contraindications to medical thoracoscopy like:

Inability to tolerate lateral decubitus position Unstable cardiovascular or hemodynamic status Presence of severe, uncorrectable hypoxemia despite oxygen therapy Bleeding diathesis Refractory cough Drug Hypersensitivity Reduced general health status with short suspected survival

* Refusal to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2020-11-11 (Actual); Primary Completion 2021-01-10 (Estimated); Study Completion 2021-01-15 (Estimated)

PRIMARY OUTCOMES:
Comparison between pleural biopsy specimens obtained by modified cryoprobe technique and conventional rigid forceps during medical thoracoscopy in diagnosis of pleural effusion regarding size of the obtained pleural biopsies. | Immediately after ending the procedure
  Size of the pleural biopsies obtained by both procedures will be compared in millimeters
Comparison between pleural biopsy specimens obtained by modified cryoprobe technique and conventional rigid forceps during medical thoracoscopy in diagnosis of pleural effusion regarding depth of the obtained pleural biopsies. | 1 week
  Depth of the pleural biopsies obtained by both procedures will be compared by "grading of fat cells" Grading will be as follows: if there will be no presence of fat cells, this will be marked as negative and if less than 5% of the biopsy will be marked as + and if 5-25% of the biopsy will be marked as ++ and if more than 25% it will take +++ in both limbs of the cryo and forceps techniques.
Comparison between pleural biopsy specimens obtained by modified cryoprobe technique and conventional rigid forceps during medical thoracoscopy in diagnosis of pleural effusion regarding integrity of the obtained pleural biopsies. | 1 week
  Integrity of the pleural biopsies obtained by both procedures will be compared by percentage of "crushed cells."" Grading will be as follows: if there will be no presence of crushed cells, this will be marked as negative and if less than 5% of the biopsy will be marked as + and if 5-25% of the biopsy will be marked as ++ and if more than 25% it will take +++ in both limbs of the cryo and forceps techniques.

SECONDARY OUTCOMES:
Safety of the procedure of thoracoscopic pleural biopsies | During the period of hospital stay
  Recording of any complications during the period of hospital stay.

CONTACTS AND LOCATIONS:
Overall Officials: Ayman I Baess, PhD, Principal Investigator — Associate Professor of Chest diseases, Alexandria University
Locations (1):
- Chest Department, Alexandria Faculty of Medicine, Alexandria, Egypt

IPD SHARING:
Plan to Share IPD: No
Data should be confirmed in larger, multi-sites studies.